CLINICAL TRIAL: NCT02406560
Title: A Phase 1, Open-label, Randomized, Crossover, Oral, Single Dose Study To Estimate The Relative Bioavailability Of Pf-06291826 (Tafamidis) Following Administration Of A Tafamidis Free Acid Tablet Formulation In Healthy Subjects Under Fasted And Fed Conditions
Brief Title: A Study Comparing The Amounts of Tafamidis In The Blood With Or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461050; 2015-000706-19 (EudraCT Number)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 tablets of 12.2 mg tafamdis free acid (Experimental)
  Interventions: Drug: tafamidis
- 4 tablets of 12.2 mg tafamidis free acid (Experimental)
  Interventions: Drug: tafamidis
- 5 tablets of 12.2 mg tafamidis free acid (Experimental)
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — fasted
  Arms: 4 tablets of 12.2 mg tafamdis free acid
Drug: tafamidis — high fat meal
  Arms: 4 tablets of 12.2 mg tafamidis free acid
Drug: tafamidis
  Other Names: fasted
  Arms: 5 tablets of 12.2 mg tafamidis free acid

SUMMARY:
Each subject will be given tafamidis after either a high fat meal or while fasted. After swallowing tafamidis, tafamidis blood concentrations will be measured periodically for one week. After about 14 days, subjects will take either a different dose of tafamidis or the same dose under the opposite meal condition. Tafamidis concentrations from the three different conditions will be compared to determine if they are approximately the same.

ELIGIBILITY:
Inclusion Criteria: - Healthy males or females of non-child bearing potential. - Body Mass Index (BMI) of 17.5 to 30.5 and total body weight more than 50 kg (110 lbs).

Exclusion Criteria: - Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic). - Use of prescription or nonprescription drugs supplements within 7 days prior to 7 days of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) | 168 hours
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Maximum Observed Plasma Concentration (Cmax) | 168 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 168 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 168 hours
Plasma Decay Half-Life (t1/2) | 168 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium